CLINICAL TRIAL: NCT00453908
Title: Does Alfuzosin OD vs. Placebo in Male Patients Facilitate Spontaneous Voiding During Clean Intermittent Self-Catheterization Following Acute Urinary Retention?
Brief Title: Alfuzosin Versus Placebo in Acute Urinary Retention
Acronym: ALF-RIK
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was early terminated due to slow and difficult recruitment
Sponsor: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: L_9397
Record Dates: First submitted 2007-03-28; First posted 2007-03-29 (Estimated); Last update posted 2007-08-20 (Estimated); Status verified 2007-08

CONDITIONS: Urinary Retention
MeSH Terms: conditions — Urinary Retention | interventions — alfuzosin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Alfuzosin

SUMMARY:
The primary objective of the study is to investigate if 14 days of treatment with Alfuzosin compared to placebo, will increase the number of patients with satisfying spontaneous voiding after acute urinary retention treated with Clean Self-Catheterization.

Furthermore is investigated the safety of the medical treatment and self-catheterization.

ELIGIBILITY:
Inclusion Criteria:

* Men with acute urinary retention and catheterized
* Benign hypertrophia of prostate
* Patient is diagnosed in Emergency room or at a acute hospitalization

Exclusion Criteria:

* Known prostate cancer
* Prior urinary retention within 30 days
* Urinary retention occurring in relation to surgery
* Blood in urine
* Difficult or impossible catheterization
* Fever > 38 degree Celsius
* Decreased kidney function
* Permanent catheter > 14 days
* Treatment with alfa 1 blocker within 30 days
* Meeting contraindications to treatment with Alfuzosin
* Treatment with other drugs for urinary problems

The above information is not intended to contain all considerations relevant to a patients potential participation in a clinical trial.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160
Dates: Start 2004-05

PRIMARY OUTCOMES:
Number of patients with satisfying spontaneous voiding after 14 days measured by bladder scan at day 14.

SECONDARY OUTCOMES:
Number of days until termination of self catheterization
Number of patients with urinary infection requiring treatment
Pressure of voiding, volume of voiding, residual urine after voiding, measured by urine culture and bladder scan at day 14.

CONTACTS AND LOCATIONS:
Overall Officials: Henning Andersen, MD, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Hoersholm, Denmark